CLINICAL TRIAL: NCT06286696
Title: Point-of-care Ultrasound of Optic Nerve Sheath Diameter in Suspected Hypertensive Emergency
Brief Title: Optic Nerve Sheath Diameter in Hypertensive Emergency
Acronym: OpticUS
Status: Not yet recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Tessa Mulder, Principal Investigator, Leiden University Medical Center
Other Study IDs: NL84914.058.23
Record Dates: First submitted 2024-01-30; First posted 2024-02-29 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hypertensive Emergency; Papilledema; Hypertension
MeSH Terms: conditions — Hypertensive Crisis; Papilledema; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optic Nerve Sheath Diameter — Point of care ultrasonography of the optic nerve sheath diameter

SUMMARY:
This prospective observational study investigates the potential of point-of-care ultrasonography of the optic nerve sheath diameter (ONSD) to rule out papilledema in patients with suspected hypertensive emergency. The primary focus is on assessing ONSD sensitivity in identifying papilledema (hypertensive retinopathy grade 4), while secondary endpoints include hypertensive retinopathy grade 3, hypertensive encephalopathy, and the need for intravenous rapid-acting medications to lower elevated blood pressure. This study aims to determine the diagnostic characteristics of this procedure for the diagnosis of hypertensive retinopathy, thus assessing its potential as a screening tool to rule out hypertensive retinopathy by the acute internal medicine doctor.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Any patient presenting to the emergency department (ED) with suspected hypertensive emergency i.e.: blood pressure of > 200 millimetres of mercury (mmHg) systolic and/or > 120 mmHg diastolic

Exclusion Criteria:

* Patients with preexisting optic nerve head changes such as glaucoma, pre-existing retinal artery/vein occlusions or any other condition that makes assessment of the fundi impossible.
* Primary neurological cause of hypertension: ischemic cerebrovascular incident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with suspected hypertensive emergency.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Papilledema | 2 years
  Sensitivity of ONSD > 5mm for diagnosis of papilledema

SECONDARY OUTCOMES:
Hypertensive retinopathy grade 3 & 4 combined | 2 years
  Sensitivity/specificity of the ONSD for hypertensive retinopathy grade 3 & 4 combined
Hypertensive encephalopathy | 2 years
  Sensitivity/specificity of the ONSD for hypertensive encephalopathy
Rapid acting medications administered intravenously to lower the elevated blood pressure | 2 years
  Sensitivity/specificity of the ONSD for the need for rapid acting medications administered intravenously to lower the elevated blood pressure
Presence of a bulging optic nerve disc and/or crescent sign found by ultrasonography of the optic nerve | 2 years
  Diagnostic characteristics for the presence of a bulging optic nerve disc and/or crescent sign for above mentioned diagnoses (papilledema, hypertensive retinopathy grade 3&4 combined, hypertensive encephalopathy, need for rapid acting intravenous medications to lower elevated bloodpressure).

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Mulder, MD, Principal Investigator — Leiden University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided